CLINICAL TRIAL: NCT03299504
Title: Factors Predicting Success in Lung Transplant Recipients Who Have Participated in the COLTT Program (Daily Intensive Post-hospitalization Rehabilitation): A Retrospective Review
Brief Title: Factors Predicting Success in Lung Transplant Recipients Who Have Undergone Intensive Post-operative Rehabilitation
Status: Completed | Type: Observational
Sponsor: Indiana University Health Methodist Hospital (Other)
Responsible Party: Principal Investigator, Christen DiPerna, Dedicated Physical Therapist, Indiana University Health Methodist Hospital
Other Study IDs: RCS1
Record Dates: First submitted 2017-09-08; First posted 2017-10-03 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Lung Transplant
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise — 5 days per week, 2.5 hours per day strength, balance and endurance training on an outpatient basis

SUMMARY:
This is a retrospective review of the COLTT program outcomes and factors that predict recovery of functional status after lung transplantation.

DETAILED DESCRIPTION:
The Center of Life for Thoracic Transplant (COLTT) program is a daily (5 days per week) intensive rehabilitation program for patients who have undergone lung transplant. Patients are enrolled in COLTT as part of standard care after hospital discharge. This study is a retrospective review of seventy patients that measures the efficacy of the COLTT program and establishes predictors of patient success.This study will also measure the effect of functional outcomes on hospital readmission post COLTT discharge.

ELIGIBILITY:
Inclusion Criteria:

* All patients who completed the COLTT program from May, 2016 to July, 2017.

Exclusion Criteria:

* Any COLTT patients who were not new lung transplant recipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung transplant recipients at IU Health Methodist Hospital. As part of standard care, all patients who survive to hospital discharge are referred by transplant pulmonologists to the COLTT program.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Time to reach program goals (days) | Through study completion, an average of 4 weeks
  The number of days in the COLTT program required to reach program goals ( see secondary outcomes measures)

SECONDARY OUTCOMES:
Gait speed (mph, % expected) | Through study completion, an average of 4 weeks
  Gait speed (walking speed) is measured daily on a oval track
Single leg stance performance (seconds, % expected) | Through study completion, an average of 4 weeks
  The test result of a single leg stance test. Patients stand with hands on their hips, raise one leg off the ground and hold it for as long as possible.
One-minute sit to stand performance (number, % expected) | Through study completion, an average of 4 weeks
  The test result of a one-minute sit to stand test. Patients stand/sit from a chair as many times as they can in one minute.
Six minute walk distance (feet, % expected) | Through study completion, an average of 4 weeks
  The test result of a six-minute walk test, a field test of exercise capacity

OTHER OUTCOMES:
Hospital readmission | 6 months
  Measured as number of hospital readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wickerson L, Rozenberg D, Janaudis-Ferreira T, Deliva R, Lo V, Beauchamp G, Helm D, Gottesman C, Mendes P, Vieira L, Herridge M, Singer LG, Mathur S. Physical rehabilitation for lung transplant candidates and recipients: An evidence-informed clinical approach. World J Transplant. 2016 Sep 24;6(3):517-31. doi: 10.5500/wjt.v6.i3.517. PMID 27683630
- [Background] Langer D, Burtin C, Schepers L, Ivanova A, Verleden G, Decramer M, Troosters T, Gosselink R. Exercise training after lung transplantation improves participation in daily activity: a randomized controlled trial. Am J Transplant. 2012 Jun;12(6):1584-92. doi: 10.1111/j.1600-6143.2012.04000.x. Epub 2012 Mar 5. PMID 22390625
- [Background] Walsh JR, Chambers DC, Davis RJ, Morris NR, Seale HE, Yerkovich ST, Hopkins PM. Impaired exercise capacity after lung transplantation is related to delayed recovery of muscle strength. Clin Transplant. 2013 Jul-Aug;27(4):E504-11. doi: 10.1111/ctr.12163. Epub 2013 Jul 2. PMID 23815281
- [Background] Strassmann A, Steurer-Stey C, Lana KD, Zoller M, Turk AJ, Suter P, Puhan MA. Population-based reference values for the 1-min sit-to-stand test. Int J Public Health. 2013 Dec;58(6):949-53. doi: 10.1007/s00038-013-0504-z. Epub 2013 Aug 24. PMID 23974352
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Middleton A, Fritz SL, Lusardi M. Walking speed: the functional vital sign. J Aging Phys Act. 2015 Apr;23(2):314-22. doi: 10.1123/japa.2013-0236. Epub 2014 May 2. PMID 24812254
- [Background] Dierich M, Tecklenburg A, Fuehner T, Tegtbur U, Welte T, Haverich A, Warnecke G, Gottlieb J. The influence of clinical course after lung transplantation on rehabilitation success. Transpl Int. 2013 Mar;26(3):322-30. doi: 10.1111/tri.12048. Epub 2013 Jan 7. PMID 23294442